CLINICAL TRIAL: NCT05056909
Title: Kidney AI-enabled Care Transformation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding refused
Sponsor: Medical University of Graz (Other)
Collaborators: Fraunhofer Institut für Arbeitswirtschaft und Organisation (Unknown); Empirica (Unknown); IN-JET APS (Unknown); CNET Svenska AB (Unknown); XIGME (Unknown); European ESKD Patients' Federation (Unknown); Catholic University of the Sacred Heart (Other); University of Manchester (Other); Università degli studi di Verona (Unknown); University of Leeds (Other); Roche Diagnostics International AG (Industry); Federación Nacional ALCER (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kidney ACTion
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; End stage kidney disease; Artificial intelligence; Patient engagement; Progression
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Patient Participation; Disease Progression | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): CKD care, as routinely provided in the respective nephrology outpatient clinic.
  Interventions: Other: Standard of care
- Intervention (Experimental): standard of care + Kidney ACTion AI-supported software for chronic kidney disease care.
  Interventions: Device: Kidney ACTion

INTERVENTIONS:
Device: Kidney ACTion — AI-supported software for chronic kidney disease care
  Arms: Intervention
Other: Standard of care — Standard of care
  Arms: Standard of care

SUMMARY:
In the Kidney ACTion study, CKD (Chronic Kidney Disease) patients at increased risk of progression to ESRD (End Stage Renal Disease) will be randomly assigned to either standard of care in a specialist nephrology outpatient clinic or to receiving CKD care supported by a novel AI-supported (Artificial Intelligence) software solution.

DETAILED DESCRIPTION:
The Advancing American Kidney Health (AAKH) initiative has the goal of an ambitious 25% reduction of ESRD incidence by 2030. There is a lack of successful integrated care programs to reach this goal. The CKD population is very heterogeneous, this explains the different risk of progression to ESRD in different patients. However, Guidelines (GLs) for the treatment of CKD patients address risk factors identified in the CKD population at large. Thus, all CKD patients at the same stage receive similar treatments no matter the specific risk of developing ESRD. Up to 5.9% of Europeans have CKD stages 3-5. Treating this huge number of patients would strain health systems from both the organizational and economical point of view. It is reasonable to think that dedicating a personalized management specifically to CKD patients at high risk of progression would be cost-effective.

GLs include behavioral (e.g. lifestyle, nutrition) as well as medical (e.g. drug therapy) interventions. Although patient's engagement and empowerment play a pivotal role in successful disease treatment, there is lack of evidence on practices to foster them in CKD patients.

Kidney ACTion is a program that supports nephrologists in predicting disease progression for CKD patients and developing multidisciplinary, personalized, evidence-based treatment and care plans. Patient engagement and empowerment is a fundamental part of the program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years at the time of signing the informed consent
* Chronic kidney disease with eGFR <45 mL/min/1.73 m2 and UACR >300 mg/g creatinine (eGFR=estimated glomerular filtration rate; UACR=Urine Albumin-to-Creatinine Ratio)
* Patient is willing to comply with the study requirements for therapy during the entire study period
* Patient is capable of providing written informed consent to participate in the study

Exclusion Criteria:

* Patients with underlying renal disease likely to receive disease-specific therapy other than SoC (Standard of Care)
* Patient expected to require renal replacement therapy within less than one year from study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Urinary Albumin to Creatinine Ratio (UACR) | 1 year after start of treatment
  Urine Albumin (mg/dL) / Urine Creatinine (g/dL) = UACR in mg/g ≈ Albumin excretion in mg/day

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Kirsch, MD, Principal Investigator — Medical University of Graz
Locations (2):
- Università Cattolica del Sacre Cuore, Roma, Italy
- University of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No